CLINICAL TRIAL: NCT05039801
Title: A Phase 1 Open-Label, Dose-Escalation and Dose-Expansion Study to Investigate the Safety, Pharmacokinetics, and Anti-Tumor Activity of IACS-6274 as Monotherapy and in Combination in Patients With Advanced Solid Tumors
Brief Title: IACS-6274 With or Without Bevacizumab and Paclitaxel for the Treatment of Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0265; NCI-2021-09063 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2021-0265 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-09-01; First posted 2021-09-10 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Advanced Endometrial Carcinoma; Advanced Head and Neck Squamous Cell Carcinoma; Advanced Malignant Solid Neoplasm; Advanced Melanoma; Advanced Ovarian Clear Cell Adenocarcinoma; Chondrosarcoma; Clinical Stage III Cutaneous Melanoma AJCC v8; Clinical Stage IV Cutaneous Melanoma AJCC v8; Pathologic Stage III Cutaneous Melanoma AJCC v8; Pathologic Stage IIIA Cutaneous Melanoma AJCC v8; Pathologic Stage IIIB Cutaneous Melanoma AJCC v8; Pathologic Stage IIIC Cutaneous Melanoma AJCC v8; Pathologic Stage IIID Cutaneous Melanoma AJCC v8; Pathologic Stage IV Cutaneous Melanoma AJCC v8; Recurrent Ovarian High Grade Serous Adenocarcinoma; Refractory Endometrial Carcinoma; Refractory Head and Neck Squamous Cell Carcinoma; Refractory Melanoma; Refractory Ovarian Clear Cell Adenocarcinoma; Refractory Ovarian High Grade Serous Adenocarcinoma; Stage III Ovarian Cancer AJCC v8; Stage III Uterine Corpus Cancer AJCC v8; Stage IIIA Ovarian Cancer AJCC v8; Stage IIIA Uterine Corpus Cancer AJCC v8; Stage IIIA1 Ovarian Cancer AJCC v8; Stage IIIA2 Ovarian Cancer AJCC v8; Stage IIIB Ovarian Cancer AJCC v8; Stage IIIB Uterine Corpus Cancer AJCC v8; Stage IIIC Ovarian Cancer AJCC v8; Stage IIIC Uterine Corpus Cancer AJCC v8; Stage IIIC1 Uterine Corpus Cancer AJCC v8; Stage IIIC2 Uterine Corpus Cancer AJCC v8; Stage IV Ovarian Cancer AJCC v8; Stage IV Uterine Corpus Cancer AJCC v8; Stage IVA Ovarian Cancer AJCC v8; Stage IVA Uterine Corpus Cancer AJCC v8; Stage IVB Ovarian Cancer AJCC v8; Stage IVB Uterine Corpus Cancer AJCC v8
MeSH Terms: conditions — Chondrosarcoma; Endometrial Neoplasms; Squamous Cell Carcinoma of Head and Neck; Melanoma; Ovarian Neoplasms | interventions — Bevacizumab; Immunoglobulin G; Disulfides; Paclitaxel; Taxes; capivasertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A (IACS-6274) (Experimental): Patients receive IACS-6274 PO throughout the study.
  Interventions: Drug: Glutaminase-1 Inhibitor IACS-6274
- Part B (IACS-6274, bevacizumab, paclitaxel) (Experimental): Patients receive IACS-6274 PO, paclitaxel IV, and bevacizumab IV throughout the study.
  Interventions: Biological: Bevacizumab; Drug: Glutaminase-1 Inhibitor IACS-6274; Drug: Paclitaxel
- PART C: (IACS-6274) with capivasertib (Experimental): Patients receive IACS-627 PO, with capivasertib PO throughout the study.
  Interventions: Drug: Glutaminase-1 Inhibitor IACS-6274; Drug: Capivasertib

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: ABP 215; Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF Monoclonal Antibody SIBP04; Anti-VEGF rhuMAb; Avastin; Bevacizumab awwb; Bevacizumab Biosimilar ABP 215; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar CT-P16; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar GB-222; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar Mvasi; Bevacizumab Biosimilar MYL-1402O; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar QL1101; Bevacizumab Biosimilar RPH-001; Bevacizumab Biosimilar SCT501; Bevacizumab Biosimilar Zirabev; Bevacizumab-awwb; Bevacizumab-bvzr; BP102; BP102 Biosimilar; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Mvasi; MYL-1402O; QL1101; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501; SIBP 04; SIBP-04; SIBP04; Zirabev
  Arms: Part B (IACS-6274, bevacizumab, paclitaxel)
Drug: Glutaminase-1 Inhibitor IACS-6274 — Given by PO
  Other Names: GLS1 Inhibitor IACS-6274; IACS 6274; IACS-6274; IACS6274; IPN 60090; IPN-60090; IPN60090
Drug: Paclitaxel — Given by IV (vein)
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
  Arms: Part B (IACS-6274, bevacizumab, paclitaxel)
Drug: Capivasertib — Given by PO
  Other Names: AZD5363
  Arms: PART C: (IACS-6274) with capivasertib

SUMMARY:
To find the highest tolerable dose of IACS-6274 that can be given alone, in combination with bevacizumab and paclitaxel, or in combination with capivasertib to patients who have solid tumors. The safety and tolerability of the study drug(s) will also be studied.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety and tolerability of oral glutaminase inhibitor IPN60090 (IACS-6274) as monotherapy (Part A) and in combination therapy with bevacizumab and weekly paclitaxel (Part B) and in combination with capivasertib (Part C)

II. To determine the maximum tolerated dose (MTD) and the recommended phase 2 dose (RP2D) of IACS-6274 in combination with bevacizumab and weekly paclitaxel (Part B). and of the combination of IACS-6274 and capivasertib (Part C). (For Dose Escalation Only)

SECONDARY OBJECTIVES:

I. To assess the preliminary antitumor activity of IACS-6274 as monotherapy (Part A) in patients with or without biomarker selected tumor types.

II. To assess the preliminary antitumor activity of IACS-6274 in the combination with bevacizumab and weekly paclitaxel (Part B) in patients with recurrent platinum-resistant ovarian cancer and in combination with capivasertib (Part C) for all solid tumors.

III. To characterize the pharmacokinetics (PK) profile of IACS-6274 as a monotherapy (Part A) and in combination with bevacizumab and weekly paclitaxel (Part B) in the combination with capivasertib (Part C). To evaluate biomarkers of patient stratification and correlate them with clinical outcome.

EXPLORATORY OBJECTIVE:

I. To collect biobank samples for potential future analysis of biomarkers (optional, informed consent required).

OUTLINE: This is a dose-escalation study of IACS-6274 followed by a dose-expansion study. Patients are assigned to 1 of 2 parts.

PART A: Patients receive IACS-6274 orally (PO) throughout the study.

PART B: Patients receive IACS-6274 PO, paclitaxel intravenously (IV), and bevacizumab IV throughout the study.

PART C: Patients receive IACS-627 PO, with capivasertib PO throughout the study.

ELIGIBILITY:
Inclusion Criteria All Parts

1. Provision of written informed consent prior to any study related procedures and compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
2. Male or female patients ≥18 years of age at the time of study entry who agree to participate by giving written informed consent prior to participation in any study related activities.
3. Histologically or cytologically confirmed advanced solid tumors, specifically:

   Dose Escalation for Part A may include:

   Patients with tumors harboring actionable KEAP1/NFE2L2/STK11/NF1 mutations Patients with low ASNS expression levels (HGSOC or endometrial cancer) Patients who had immunotherapy (IO) melanoma (Minimum treatment duration of prior PD-1 or PD-L1-containing regimen of 12 weeks [or equivalent of 2 response evaluations]).

   Patients with post-platinum HNSCC Patients with chondrosarcoma Patients with ARID1A mutant clear cell ovarian cancer

   Dose Escalation for Part B may include:

   Confirmed recurrent high-grade non-mucinous ovarian cancer that is platinum-resistant, defined as disease relapse within a platinum-free interval (PFI, or the time elapsed from the last date of platinum dose until PD) of < 6 months, and with less than 5 prior therapies

   Dose Expansion for Part B limited to:

   Confirmed recurrent high-grade non-mucinous ovarian cancer with low ASNS expression levels that is platinum-resistant, defined as disease relapse within a PFI of < 6 months, and with less than 5 prior therapies.

   Dose Escalation for Part C may include:

   Patients with tumors harboring actionable KEAP1/NFE2L2 mutations Patients with tumors harboring PIK3CA hotspot mutations, activating AKT mutations, and inactivating PTEN mutations (irrespective of KEAP1/NFE2L2 mutations) Patients with low ASNS expression levels (HGSOC)

   Dose Expansion for Part C limited to:

   Patients with NSCLC with actionable KEAP1/NFE2L2 mutations Patients with HGSOClow ASNS expression levels (irrespective of biomarker status for KEAP1/NFE2L2)
4. Patients must have received at least one line of therapy for advanced stage disease and be refractory or ineligible to available existing therapy(ies) known to provide clinical benefit for their condition.
5. Prior treatment with chemotherapy, radiotherapy, immunotherapy or any investigational therapies must have been completed at least 3 weeks or at least five half lives, whichever is shorter, before the study drug administration, and all AEs (excluding alopecia and peripheral neuropathy) have either returned to ≤Grade 1 or stabilized. Patients with concurrent use of hormonal therapy for non-cancer related conditions (e.g., hormone replacement therapy) are allowed.
6. Fresh and/or archival tumor tissue from a biopsy obtained between the completion of the most recent line of treatment until study entry must be available for mutation and biomarker analysis. If available, archival tumor tissue from the time of initial diagnosis or the most recent biopsy (archival and/or fresh) will be collected. For ovarian cancer patients, a fresh biopsy must be collected in addition to archival tumor tissue. NOTE: No fresh tumor tissue will be required if a previous biopsy detected the selected mutations for each cohort. In all cases, procedures to obtain fresh tumor tissue should not put the patient at undue risk, and should only be performed if the risk is minimal (no greater than 2% risk of serious or severe complications).
7. Patients must have at least 1 lesion (measurable and/or non-measurable) that can be accurately assessed at baseline by CT or MRI and is suitable for repeated assessments.
8. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤1 with no deterioration over the previous 2 weeks prior to baseline or day of first dosing.
9. Adequate organ function as indicated by the following laboratory values:

   Absolute neutrophil count (ANC) ≥1.0×109/L Platelets ≥100×109/L Hemoglobin ≥9.0 g/dL (>5.59 mmol/L) Creatinine clearance (CrCl) >50 mL/min. Actual body weight should be used for calculating creatinine clearance using the Cockroft Gault equation (except for patients with body mass index >30 kg/m2 when the lean body weight should be used, and without the need for chronic dialysis therapy).

   Serum total bilirubin ≤1.5×ULN (with the exception of patients with known thalassemia minor mutations or Gilbert's syndrome: serum total bilirubin must be <3×ULN in these patients) Aspartate aminotransferase (serum glutamic oxaloacetic transaminase) and alanine aminotransferase (serum glutamic pyruvic transaminase) ≤2.5×ULN or ≤5×ULN for patients with liver metastases)
10. Adequate cardiac function with a left ventricular ejection fraction ≥50%
11. Female patients of non childbearing potential, who are physiologically incapable of becoming pregnant, are eligible to enter and participate in the study if they:

    have had a hysterectomy, OR have had a bilateral oophorectomy, OR have had a bilateral salpingectomy, OR is postmenopausal (total cessation of menses for ≥2 years, or follicle stimulating hormone ≥50 IU/L).
12. Female patients of childbearing potential, who are not post-menopausal or surgically sterile and intent to be sexually active with a non-sterile male partner, are required to use one form of highly effective contraception combined with a barrier method (male condom, female condom, cervical cap, diaphragm with spermicide, or contraceptive sponge with spermicide) of contraception starting before entering the study and until 4 weeks after the last dose of treatment.

    Highly effective non-hormonal contraceptive methods that are acceptable include:

    Total/true abstinence*** for the total duration of the study treatment and for at least 1 month after the last dose of study treatment. Periodic abstinence using methods such as calendar ovulation, symptothermal, post ovulation methods, declaration of abstinence solely for the duration of a trial, or withdrawal are not acceptable methods of contraception.

    Having a vasectomized sexual partner, who received post-vasectomy confirmation of azoospermia, combined with a barrier method as described above.

    Bilateral tubal occlusion combined with a barrier method as described above. Intrauterine device with copper banded coils, combined with a barrier method as described above.

    Highly effective hormonal contraceptive methods that are acceptable include:

    Combined oral pill contraception (normal and low-dose oral pills, or progesterone-based oral pills using desogestrel) combined with a barrier method as described above. NOTE: cerazette is currently the only highly efficacious progesterone-based pill available.

    Injection (e.g., medroxyprogesterone) combined with a barrier method as described above.

    Patch (e.g., norelgestromin or ethinyl estradiol transdermal system) combined with a barrier method as described above.

    Implants (etonorgestrel-releasing) combined with a barrier method as described above.

    Intravaginal device (e.g., ethinyl estradiol- or etonogestrel-releasing) combined with a barrier method as described above.

    Intrauterine system (levonorgestrel-releasing) combined with a barrier method as described above.

    In addition to the to use one form of highly effective contraception combined with a barrier method, female patients of childbearing potential must have a negative serum pregnancy test at screening (within 7 days of the start of treatment) and must not be breastfeeding.
13. Non-sterile men, who are not sexually abstinent and intend to be sexually active with a woman of childbearing potential, must use a condom from the start of the trial and until 16 weeks after the last dose of treatment, or must practice total abstinence*** for the total duration of the study treatment and at least 3 months after the last dose of study treatment. Periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of contraception. Female partners of childbearing potential should consider the use of at least one contraception method describe above. If the female partner is pregnant, male participants should use a condom plus spermicide.

    * Total/true abstinence is defined as a patient who refrains from any form of sexual intercourse, and this is in line with their usual and/or preferred lifestyle.

Exclusion Criteria All Parts

1. Prior malignancy within the previous 2 years except for locally curable cancers that have been cured, such as basal or squamous cell skin cancer, or carcinoma in situ of the cervix, breast or bladder.
2. Known primary central malignancy or symptomatic central nervous system metastasis(es).

   Note: Patients with stable, previously treated brain metastases may participate if neurologic symptoms have resolved, patients have been off steroids (at least 7 days for Part A and Part B, and at least 4 weeks for Part C), and there is no evidence of disease progression by imaging for at least 2 weeks before the first dose of study treatment.
3. Uncontrolled, significant intercurrent or recent illness including, but not limited to, the following cardiac conditions:

   1. Any unstable cardiac arrhythmia within 6 months prior to enrolment
   2. Prolongation of the Fridericia corrected QT (QTcF) interval defined as >450 ms for males and >470 ms for females
   3. History of any of the following cardiovascular conditions within 6 months of enrolment:

      * cardiac angioplasty or stenting, myocardial infarction, unstable angina, coronary artery bypass graft surgery, symptomatic peripheral vascular disease, class III or IV congestive heart failure, as defined by the New York Heart Association.
4. Major surgical intervention within 28 days before study drug administration, or an anticipated need for major surgery during the study.
5. Significant acute or chronic infections.
6. Any psychiatric condition that would prohibit the understanding or rendering of informed consent.
7. Treatment with strong cytochrome P450 subtype 3A4 (CYP3A4) inducers and inhibitors (including grapefruit juice) within 2 weeks of the first dose of study drug NOTE: patients must have stopped taking St. John's Wort 3 weeks prior to the start of treatment and stopped taking enzalutamide 4 weeks prior to the start of treatment.
8. Treatment with strong CYP450 subtype 2D6 (CYP2D6) inhibitors or sensitive CYP3A4 substrates within 7 days of the first dose of study drug.
9. Radiotherapy within 4 weeks prior to the start of study drug. Palliative radiotherapy for symptomatic control is acceptable if completed at least 2 weeks prior to study drug administration and no additional radiotherapy for the same lesion is planned.
10. Underlying medical conditions (such as severe or uncontrolled systemic diseases, including uncontrolled hypertension, renal transplant and active bleeding diseases), for which in the investigator's opinion will make the administration of study drug hazardous or obscure the interpretation of toxicity determination or AEs.
11. History of allergic reactions attributed to compounds of similar chemical or biological composition to any of the compounds in the study.
12. Known history of alcohol or drug abuse.
13. Legal incapacity or limited legal capacity.
14. Inability to swallow oral medications (capsules and tablets) without chewing, breaking, crushing, opening or otherwise altering the product formulation. Patients should not have gastrointestinal illnesses (such as refractory nausea and vomiting, chronic gastrointestinal disease or previous significant bowel resection that would preclude adequate absorption, distribution, metabolism, or excretionof IACS-6274 and capivasertib, which are oral agents.
15. Patients unwilling to comply with protocol requirements related to the assigned part.
16. Any other disease, physical examination finding, or clinical laboratory finding that, in the investigator's opinion, gives reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug, may affect the interpretation of the results, render the patient at high risk from treatment complications or interferes with obtaining informed consent.

Part B Specific Exclusion Criteria (B1) Known severe hypersensitivity reactions to monoclonal antibodies, any history of anaphylaxis, or uncontrolled asthma (that is, three or more features of partially controlled asthma).

(B2) Patient has a known hypersensitivity to paclitaxel or bevacizumab components or excipients.

(B3) Patient has a history of bowel obstruction, including sub-occlusive disease, related to the underlying disease and history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscesses. Evidence of recto-sigmoid involvement by pelvic examination or bowel involvement on CT scan or clinical symptoms of bowel obstruction.

(B4) Patient has proteinuria as demonstrated by urine protein:creatinine ratio ≥1.0 at screening or urine dipstick for proteinuria ≥2 (patients discovered to have ≥2 proteinuria on dipstick at baseline should undergo 24-hour urine collection and must demonstrate <2 g of protein in 24 hours to be eligible).

(B5) Patient is at increased bleeding risk due to concurrent conditions (e.g., major injuries or surgery within the past 28 days prior to start of study treatment, history of hemorrhagic stroke, transient ischemic attack, subarachnoid hemorrhage, or clinically significant hemorrhage within the past 3 months).

(B6) Patient has clinically significant cardiovascular disease (e.g., significant cardiac conduction abnormalities, uncontrolled hypertension, myocardial infarction, cardiac arrhythmia or unstable angina, New York Heart Association Grade 2 or greater congestive heart failure, serious cardiac arrhythmia requiring medication, Grade 2 or greater peripheral vascular disease, and history of cerebrovascular accident [CVA]) within 6 months of enrollment. (B7) Patient has pre-existing peripheral neuropathy that is Grade ≥2 by Common Terminology Criteria for Adverse Events (CTCAE) version 4 criteria.

(B8) Patient requires paracentesis 2 weeks prior to trial enrolment. Part C Specific Exclusion Criteria (C1) History of another primary malignancy, except for a malignancy treated with curative intent, with no known active disease ≥5 years before the first dose of treatment, with low potential risk for recurrence. Exceptions include basal cell carcinoma of the skin and squamous cell carcinoma of the skin that has undergone potentially curative therapy.

(C2) Patient has a known hypersensitivity to capivasertib components or any excipients of the product.

(C3) Clinically significant abnormalities of glucose metabolism as defined by any of the following: Diagnosis of diabetes mellitus type I or II (irrespective of management), Glycosylated haemoglobin (HbA1c) >8% (64 mmol/mol) (C4) Patients with evidence of severe or uncontrolled systemic liver disease including severe hepatic impairment, or abnormal liver enzymes at screening (AST or ALT >2.5 x ULN; total bilirubin >1.5 x ULN).

(C5) Patients with elevated alkaline phosphatase (ALP) can be enrolled if the abnormal value is due to the presence of bone metastasis, but liver function is considered adequate according to the principal investigator.

(C6) Patients with persistent toxicities (Grade ≥2 by Common Terminology Criteria for Adverse Events (CTCAE) version 4) caused by previous anticancer therapy, excluding alopecia. Participants with irreversible toxicity that is not reasonably expected to be exacerbated by study treatment may be included after consultation with the sponsor and the study physician.

(C7) Patients with spinal cord compression or leptomeningeal disease not requiring steroids for at least 4 weeks prior to start of study intervention.

(C8) Patients with clinically significant cardiovascular disease including, but not limited to, significant cardiac conduction abnormalities, uncontrolled hypertension, myocardial infarction, cardiac arrhythmia or unstable angina, New York Heart Association Grade 2 or greater congestive heart failure, serious cardiac arrhythmia requiring medication, Grade 2 or greater peripheral vascular disease, and history of cerebrovascular accident [CVA]) within 6 months of enrollment. In addition, patients will be excluded based on the study physician's judgment of the following criteria:

* Mean resting corrected QT interval >470ms, obtained from triplicate ECGs performed at screening.
* Medical history significant for arrhythmia that is symptomatic or requires treatment (CTCAE Grade 3), symptomatic or uncontrolled atrial fibrillation regardless of treatment, or asymptomatic sustained ventricular tachycardia. Participants with atrial fibrillation controlled by medication or arrhythmias controlled by pacemakers may be included based on the study physician's judgment.
* Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalemia of Grade ≥1, potential for Torsades de Pointes, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age in first-degree relative, history of QT prolongation associated with other medications that required discontinuation of the medication.
* Experience of any of the following procedures or conditions in the preceding 6 months: coronary artery bypass graft, angioplasty, vascular stent, myocardial infarction, angina pectoris, congestive heart failure New York Heart Association Grade ≥2.
* Uncontrolled hypotension: SBP <90 mmHg and/or DBP <50 mmHg.
* Cardiac ejection fraction outside institutional range of normal or <50% (whichever is higher) as measured by echocardiogram (or multiple-gated acquisition [MUGA] scan if an echocardiogram cannot be performed or is inconclusive).

(C9) Patients with active tuberculosis infection (clinical evaluation that may include clinical history, physical examination and radiographic findings, or tuberculosis testing in line with local practice) are excluded.

(C10) Patients with active hepatitis infection, positive hepatitis C antibody, hepatitis B virus surface antigen or hepatitis B virus core antibody, at screening are excluded.

Human immunodeficiency virus (HIV) positive patients with a viral load > 400 copies/mL and a CD4+ T-cell count of <350 cells/uL or with a history of an acquired immunodeficiency syndrome (AIDS) opportunistic infection within the past 12 months are excluded. Patients with a higher viral load or lower CD4+ count (< 350 cells/uL) may be considered for eligibility if the patient has a potentially curable malignancy or for interventions in a later stage of development that have demonstrated prior activity with a given cancer.

HIV-positive patients receiving antiretroviral therapies should be on established ART for at least four weeks before starting treatment to ensure that treatment is tolerated and that toxicities are not confused with investigational drug toxicities. HIV-positive patients receiving antiretroviral therapies that are strong CYP3A4/5 inhibitors/ inducers or sensitive substrates of CYP3A4 will be excluded due to the potential for drug-drug interaction with capivasertib.

(C12) Patients who are undergoing any concurrent anticancer treatment or any concomitant medication that may interfere with the study drugs according to local clinical guidelines are excluded.

(C13) Patients who received palliative radiotherapy within 2 weeks prior to the start of study treatment; or radiotherapy to more than 30% of the bone marrow within 4 weeks before the start of study treatment are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2021-09-09 (Actual); Primary Completion 2026-05-29 (Estimated); Study Completion 2026-05-29 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 90 days
  Will be assessed by the rate of dose limiting toxicities at each dose level in the dose escalation, and the rate of AEs and the rate of Grade 3 and higher AEs in the dose escalation and dose expansion. All AEs will be coded according to the latest version of Medical Dictionary for Regulatory Activities and National Cancer Institute-Common Terminology Criteria for Adverse Events version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy A Yap, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org